CLINICAL TRIAL: NCT03888677
Title: SBG 2000-1. Individually Dose-adjusted FEC Compared to Standard FEC as Adjuvant Chemotherapy for Node Positive or High-risk Node Negative Breast Cancer. A Randomized Study by the Scandinavian Breast Group
Brief Title: Dose-adjusted Adjuvant FEC Compared to Standard FEC for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henrik Lindman (Other)
Collaborators: Scandinavian Breast Group (Other); Danish Breast Cancer Cooperative Group (Other); Swedish Cancer Society (Other); Swedish Cancer Foundation (Other); Pharmacia Pharmaceutical Company (Unknown); Swedish Breast Cancer Group (Other)
Responsible Party: Sponsor-Investigator, Henrik Lindman, Senior Consultant, Ass. Professor, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBG 2000-1
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard (Active Comparator): Standard FEC (F600, E60, C600) every 3rd week.
  Interventions: Drug: 5-FU, epirubicin and cyclophosphamide
- Tailored (Experimental): Tailored FEC (F600, E75-90, C900-1200) every 3rd week.
  Interventions: Drug: 5-FU, epirubicin and cyclophosphamide
- Registered (Active Comparator): Non-randomized arm with patients with grade 3-4 leukopenia after first cycle and treated with standard FEC (F600, E60, C600) every 3rd week.
  Interventions: Drug: 5-FU, epirubicin and cyclophosphamide

INTERVENTIONS:
Drug: 5-FU, epirubicin and cyclophosphamide — Tailored dose escalation of epirubicin and cyclophosphamide.

SUMMARY:
This is an open randomized phase III study. The primary objective of this study is to compare FEC adjuvant chemotherapy in operable breast cancer given either as fixed doses calculated according to the patients surface area or with doses adjusted according to leukopenia after course one in order to achieve hematological equitoxicity. The main aim of the study is to test whether chemotherapy dosage aimed at hematological equitoxicity will improve the effect of adjuvant chemotherapy.

DETAILED DESCRIPTION:
Group A, FECStandard(standard FEC) is given 7 courses of 5-fluorouracil-epirubicin (Farmorubicin)-cyclophosphamide with doses based on the patient's surface area. Leukocyte nadir values at day 10, 12 or 13 and 15 are measured. Dose-reductions of one step according to table 8.2.1 are performed in case of leukopenic fever or grade 4 leukopenia.

Group B FECTailored(Tailored FEC) receives course one at identical doses to group A. Leukocyte nadir values at day 10,12 or 13 and 15 are measured. Doses of subsequent courses are adjusted to achieve grade 3 leukopenia (leukocyte nadir 1.0 to 2.0) in patients experiencing only grade 0 to 2 leukopenia after course one.

Dose-reductions of one step according to table 8.2.1 are performed in case of leukopenic fever or grade 4 leukopenia .

Patients achieving only grade 0-2 leukopenia at the first course will be randomized into continued treatment at standard doses (Group A) or to doses tailored to achieve grade 3 leukopenia (Group B). The primary comparisons will be made between these two groups of patients.

Patients with grade 3-4 leukopenia after the first course not be randomized but followed according to the protocol and received treatment as group A, FECStandard.

ELIGIBILITY:
Inclusion Criteria:

* Node positive or 2) High-risk node negative#
* no major cardiovascular morbidity
* female age 18-60
* ECOG/WHO performance status <1
* histologically proven invasive breast cancer
* written or oral witnessed informed consent according to the local Ethics Committee requirements
* start of adjuvant chemotherapy within 8 weeks after surgery

Exclusion Criteria:

* distant metastases (M1)
* locally advanced cancer
* nonradically operated (positive resection margins)
* pregnancy or lactation
* leukocyte count < 3.5 x109 /l
* platelets < 100 x109 /l
* other serious medical condition
* previous or concurrent malignancies at other sites, except basal cell carcinoma and carcinoma cervicis uteri in situ

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1535 (Actual)
Dates: Start 2001-02 (Actual); Primary Completion 2003-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Distant disease-free survival. | 5-10 years
  Distant disease-free survival comparing standard and tailored arm.

SECONDARY OUTCOMES:
Regio-locally relapsed disease | 5-10 years
  Regiolocal disease-free survival
Overall survival | 5-10 years
  Overall survival
Toxicity of treatment. | 5-10 years
  Adverse events
Leukopenia and correlation to prognosis in distant disease-free survival. | 5-10 years.
  Distant disease-free survival in patients groups based on nadir leukopenia after third cycle.
Effect of dose escalation of leukopenia and correlation to prognosis in distant disease-free survival. | 5-10 years.
  Comparing distant disease-free survival difference between patients randomized to tailored and dose-escalated FEC with the Group of patients with standard FEC but with similar grade of leukopenia.

IPD SHARING:
Plan to Share IPD: Yes
Sharing with EBCTCG (Early Breast Cancer Trialists' Collaborative Group).
Supporting Information: CSR
Time Frame: After 5 years.